CLINICAL TRIAL: NCT04923958
Title: Rapid Research in Diagnostics Development for TB Network (R2D2 TB Network) Study
Brief Title: Rapid Research in Diagnostics Development for TB Network
Acronym: R2D2TB Network
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University Hospital Heidelberg (Other); Christian Medical College, Vellore, India (Other); Vietnam National Lung Hospital (Unknown); De La Salle University Medical Center (Other); University of Stellenbosch (Other); Makerere University (Other); Johns Hopkins Bloomberg School of Public Health (Other); Harvard Medical School (HMS and HSDM) (Other); Stanford University (Other); Foundation for Innovative New Diagnostics, Switzerland (Other); Socios En Salud Sucursal, Peru (Other); Federal University of Mato Grosso (Other); Medical Research Council (Other Government); National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia (Other); Centre for Infectious Disease Research in Zambia (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Zankli Research Center (Unknown); University of California, Irvine (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: U01AI152087 (NIH); U01AI152087 (NIH); R01AI190419 (NIH)
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Diagnostics; Global Health
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Evaluation of various novel TB triage and diagnostic tests. (Experimental): For the novel TB triage and diagnostic tests, the investigators will conduct large-scale evaluation of design-locked tests in a cohort of adults with presumed TB, with nested feasibility/pilot studies of early and late prototype tests. The investigators aim to enroll 300-450 participants per year at each of five enrollment sites for evaluation of various novel TB triage and diagnostic tests and 50 health workers to assess test usability.
  Interventions: Diagnostic Test: Novel mycobacterial culture techniques; Diagnostic Test: Novel sputum smear microscopy techniques; Diagnostic Test: Sputum-based molecular assays; Diagnostic Test: Tongue swab-based molecular assays; Diagnostic Test: Urine LAM assays; Diagnostic Test: Blood-based host immune response assays; Diagnostic Test: Breath-based assays; Diagnostic Test: Artificial intelligence-based digital health tools; Diagnostic Test: Phage-based assays
- Evaluation of novel rDST assays (Experimental): Clinicians at participating sites will be asked to refer adult patients with rifampin-resistance identified by routine molecular testing. The investigators aim to enroll 100-200 patients per year at each of three enrollment sites for evaluation of novel rDST assays.
  Interventions: Diagnostic Test: Cartridge-based molecular assays for detecting drug resistance; Diagnostic Test: Sequencing-based assays for detecting drug resistance

INTERVENTIONS:
Diagnostic Test: Novel mycobacterial culture techniques — We will evaluate tests intended to make culture more sensitive, faster, and have less contamination.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Novel sputum smear microscopy techniques — We will evaluate new staining techniques or visualization methods to increase the sensitivity of smear microscopy.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Sputum-based molecular assays — We will evaluate semi-automated or automated molecular assays intended for use at near point of care or point of care.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Tongue swab-based molecular assays — We will evaluate semi-automated or automated molecular assays intended for use at near point of care or point of care.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Urine LAM assays — We will evaluate urine LAM assays incorporating techniques such as analyte concentration, higher sensitivity or specificity antibodies, or enhanced visualization to improve LAM detection.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Blood-based host immune response assays — We will evaluate assays measuring host immune response parameters intended for use at near point of care or point of care.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Breath-based assays — We will evaluate assays assessing volatile organic compounds or exhaled breath condensate for near point of care of point of care detection of TB.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Artificial intelligence-based digital health tools — We will evaluate AI-based algorithms evaluating images (chest x-ray, ultrasound) or sounds (cough sounds, lung sounds) including an Infrasound-to-ultrasound e-stethoscope (Level 42 AI, USA).
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Phage-based assays — We will evaluate assays using phages to lyse mycobacterial cells for detection of DNA or antigens.
  Arms: Evaluation of various novel TB triage and diagnostic tests.
Diagnostic Test: Cartridge-based molecular assays for detecting drug resistance — We will evaluate semi-automated or automated molecular assays intended for use at near point of care or point of care.
  Arms: Evaluation of novel rDST assays
Diagnostic Test: Sequencing-based assays for detecting drug resistance — We will evaluate targeted and whole genome sequencing assays.
  Arms: Evaluation of novel rDST assays

SUMMARY:
To reduce the burden of TB worldwide through more accurate, faster, simpler, and less expensive diagnosis of TB Every year, more than 3 million people with TB remain undiagnosed and 1 million die. Better diagnostics are essential to reducing the enormous burden of TB worldwide. The Rapid Research in Diagnostics Development for TB Network (R2D2 TB Network) brings together experts in TB care, technology assessment, diagnostics development, laboratory medicine, epidemiology, health economics and mathematical modeling with highly experienced clinical study sites in 10 countries.

DETAILED DESCRIPTION:
The Rapid Research in Diagnostics Development for TB Network (R2D2 TB Network) study seeks to identify and rigorously assess promising early stage tuberculosis (TB) triage, diagnostic and drug resistance tests (hereafter referred to as "novel tests") in clinical studies conducted in settings of intended use. Rapid diagnosis, identification of drug resistance and effective treatment are critical for improving patient outcomes and reducing TB transmission. However, analysis of care cascades and prevalence surveys indicate that 40-60% of patients with TB are not initiated on effective treatment.1,2 The different types of tests required to reduce this "diagnostic gap" have been described in the form of target product profiles (TPPs). The highest- priority TPPs are for: 1) a point-of-care, non-sputum biomarker-based test to facilitate rapid TB diagnosis using easily accessible samples (a biomarker-based diagnostic test) and 2) a simple, low-cost test that can be used by front-line health workers to rule-out TB (a triage test). The R2D2 TB Network study will evaluate the sensitivity and specificity of novel triage and diagnostic tests against a reference standard including sputum Xpert® MTB/RIF (Mycobacterium tuberculosis/Rifampin) Ultra and sputum mycobacterial culture. The sensitivity and specificity of rapid drug susceptibility tests (rDST) will be compared against a reference standard including culture-based phenotypic DST and whole genome sequencing (WGS) of mycobacterial DNA. In addition, the usability of novel tests will be assessed through direct observations and surveys of routine health workers.

ELIGIBILITY:
Novel TB triage and diagnostic tests:

We will include non-hospitalized adults (age ≥ 12 years) with either 1) cough ≥2 weeks' duration, a commonly accepted criterion for identifying people with presumed pulmonary TB (to facilitate standardization across sites and comparison of test performance across sub-groups or 2) risk factors for which TB screening is recommended (HIV infection, self-reported close contact, history of mining work). People with risk factors will be included if they screen positive for TB based on WHO-recommended screening tools as specified below:

Positive TB screening definitions by risk factor:

1. PLHIV (Risk Factor), CRP >5 mg/dL OR abnormal CXR (Positive TB screening definition)
2. Self-reported Close Contact (Risk Factor), abnormal CXR (Positive TB screening definition)
3. History of mining work (Risk Factor), abnormal CXR (Positive TB screening definition)

We will exclude people who:

1. completed latent or active TB treatment within the past 12 months (to increase TB prevalence and reduce false-positive results, respectively);
2. have taken any medication with anti-mycobacterial activity (including fluoroquinolones) for any reason, within 2 weeks of study entry (to reduce false-negatives);
3. reside >20km from the study site or are unwilling to return for follow-up visits; or
4. are unwilling to provide informed consent

Novel TB rDST assays:

We will include adults (age ≥12 years) who are positive for TB and RIF resistance according to routine diagnostic testing (based typically on Xpert MTB/RIF, Xpert MTB/RIF Ultra, or Hain MTBDRplus). We will exclude people who:

1. have negative or contaminated results on all baseline (i.e., enrollment) sputum cultures
2. are unable to provide at least two sputum specimens of 3 mL each within one day of enrollment
3. are unable or unwilling to provide informed consent

Assessment of the usability of novel TB tests:

We will include health workers at each clinical site who are 1) aged ≥18 years and 2) involved in routine TB testing (collecting specimens for or performing TB tests). We will exclude staff who are unwilling to provide informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26436 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2031-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 7 months
  Number of positive results for a given index test/(Total positive + negative results for a given index test) among patients with TB using the microbiological reference standard
Specificity | 7 months
  Number of negative results for a given index test/(Total positive + negative results for a given index test) among patients without TB using the microbiological reference standard

CONTACTS AND LOCATIONS:
Overall Officials: Adithya Cattamanchi, MD, Principal Investigator — University of California, San Francisco
Locations (16):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- India (3):
  - Chitoor (Christian Medical College satellite campus), Vellore
  - Christian Medical College CMC Pulmonary Outpatient Department, Vellore
  - Primary care clinics (Shalom/LCC, CHAD), Vellore
- Zankli Research Center, Abuja, Nigeria
- De La Salle Medical and Health Sciences Institute, Dasmariñas, Philippines
- South Africa (5):
  - Brooklyn Chest Hospital, Cape Town
  - Khayelitsha District Health Center, Cape Town
  - Kraaifontein Community Health Clinic, Cape Town
  - Scottsdene primary care clinic, Cape Town
  - Wallacedene primary care clinic, Cape Town
- Uganda (2):
  - Kisenyi Health Center, Kampala
  - Mulago Outpatient Department, Kampala
- Vietnam (2):
  - Hanoi Lung Hospital, Outpatient departments, Hanoi
  - National Lung Hospital, Outpatient departments, Hanoi
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho SN, Brennan PJ. Tuberculosis: diagnostics. Tuberculosis (Edinb). 2007 Aug;87 Suppl 1:S14-7. doi: 10.1016/j.tube.2007.05.001. Epub 2007 Jun 20. PMID 17584529
- [Background] World Health Organization. Global tuberculosis report Geneva, Switzerland: World Health Organization, 2015.
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Walusimbi S, Bwanga F, De Costa A, Haile M, Joloba M, Hoffner S. Meta-analysis to compare the accuracy of GeneXpert, MODS and the WHO 2007 algorithm for diagnosis of smear-negative pulmonary tuberculosis. BMC Infect Dis. 2013 Oct 30;13:507. doi: 10.1186/1471-2334-13-507. PMID 24172543
- [Background] World Health Organization. Rapid Implementation of the Xpert MTB / RIF diagnostic test. Technical and operational 'how-to' practical considerations. Geneva, Switzerland, 2011.
- [Background] Systematic Screening for Active Tuberculosis: Principles and Recommendations. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK294083/ PMID 25996015
- [Background] World Health Organization. Drug-resistant TB. https://www.who.int/tb/areas-of-work/drug-resistant-tb/en/.
- [Background] Dalton T, Cegielski P, Akksilp S, Asencios L, Campos Caoili J, Cho SN, Erokhin VV, Ershova J, Gler MT, Kazennyy BY, Kim HJ, Kliiman K, Kurbatova E, Kvasnovsky C, Leimane V, van der Walt M, Via LE, Volchenkov GV, Yagui MA, Kang H; Global PETTS Investigators; Akksilp R, Sitti W, Wattanaamornkiet W, Andreevskaya SN, Chernousova LN, Demikhova OV, Larionova EE, Smirnova TG, Vasilieva IA, Vorobyeva AV, Barry CE 3rd, Cai Y, Shamputa IC, Bayona J, Contreras C, Bonilla C, Jave O, Brand J, Lancaster J, Odendaal R, Chen MP, Diem L, Metchock B, Tan K, Taylor A, Wolfgang M, Cho E, Eum SY, Kwak HK, Lee J, Lee J, Min S, Degtyareva I, Nemtsova ES, Khorosheva T, Kyryanova EV, Egos G, Perez MT, Tupasi T, Hwang SH, Kim CK, Kim SY, Lee HJ, Kuksa L, Norvaisha I, Skenders G, Sture I, Kummik T, Kuznetsova T, Somova T, Levina K, Pariona G, Yale G, Suarez C, Valencia E, Viiklepp P. Prevalence of and risk factors for resistance to second-line drugs in people with multidrug-resistant tuberculosis in eight countries: a prospective cohort study. Lancet. 2012 Oct 20;380(9851):1406-17. doi: 10.1016/S0140-6736(12)60734-X. Epub 2012 Aug 30. PMID 22938757
- [Background] Gandhi NR, Moll A, Sturm AW, Pawinski R, Govender T, Lalloo U, Zeller K, Andrews J, Friedland G. Extensively drug-resistant tuberculosis as a cause of death in patients co-infected with tuberculosis and HIV in a rural area of South Africa. Lancet. 2006 Nov 4;368(9547):1575-80. doi: 10.1016/S0140-6736(06)69573-1. PMID 17084757
- [Background] Masjedi MR, Farnia P, Sorooch S, Pooramiri MV, Mansoori SD, Zarifi AZ, Akbarvelayati A, Hoffner S. Extensively drug-resistant tuberculosis: 2 years of surveillance in Iran. Clin Infect Dis. 2006 Oct 1;43(7):841-7. doi: 10.1086/507542. Epub 2006 Aug 21. PMID 16941364
- [Background] Prasad R, Singh A, Balasubramanian V, Gupta N. Extensively drug-resistant tuberculosis in India: Current evidence on diagnosis & management. Indian J Med Res. 2017 Mar;145(3):271-293. doi: 10.4103/ijmr.IJMR_177_16. PMID 28749390
- [Background] Yoon C, Dowdy DW, Esmail H, MacPherson P, Schumacher SG. Screening for tuberculosis: time to move beyond symptoms. Lancet Respir Med. 2019 Mar;7(3):202-204. doi: 10.1016/S2213-2600(19)30039-6. No abstract available. PMID 30823972
- [Background] Organization WH. High-priority target product profiles for new tuberculosis diagnostics: report of a consensus meeting. Geneva, Switzerland: WHO Press; 2014. p. 98.
- [Background] World Health Organization. High-priority target product profiles for new tuberculosis diagnostics: report of a consensus meeting. Geneva, Switzerland, 2014.
- [Background] UNITAID. TB Diagnostics Market in Select High-Burden Countries: Current Market and Future Opportunities for Novel Diagnostics. Geneva, Switzerland, 2015.
- [Background] Subbaraman R, Nathavitharana RR, Satyanarayana S, Pai M, Thomas BE, Chadha VK, Rade K, Swaminathan S, Mayer KH. The Tuberculosis Cascade of Care in India's Public Sector: A Systematic Review and Meta-analysis. PLoS Med. 2016 Oct 25;13(10):e1002149. doi: 10.1371/journal.pmed.1002149. eCollection 2016 Oct. PMID 27780217
- [Background] Farhat MR, Sultana R, Iartchouk O, Bozeman S, Galagan J, Sisk P, Stolte C, Nebenzahl-Guimaraes H, Jacobson K, Sloutsky A, Kaur D, Posey J, Kreiswirth BN, Kurepina N, Rigouts L, Streicher EM, Victor TC, Warren RM, van Soolingen D, Murray M. Genetic Determinants of Drug Resistance in Mycobacterium tuberculosis and Their Diagnostic Value. Am J Respir Crit Care Med. 2016 Sep 1;194(5):621-30. doi: 10.1164/rccm.201510-2091OC. PMID 26910495
- [Background] Lange C, Chesov D, Furin J, Udwadia Z, Dheda K. Revising the definition of extensively drug-resistant tuberculosis. Lancet Respir Med. 2018 Dec;6(12):893-895. doi: 10.1016/S2213-2600(18)30428-4. Epub 2018 Nov 9. No abstract available. PMID 30420247
- [Background] Makhado NA, Matabane E, Faccin M, Pincon C, Jouet A, Boutachkourt F, Goeminne L, Gaudin C, Maphalala G, Beckert P, Niemann S, Delvenne JC, Delmee M, Razwiedani L, Nchabeleng M, Supply P, de Jong BC, Andre E. Outbreak of multidrug-resistant tuberculosis in South Africa undetected by WHO-endorsed commercial tests: an observational study. Lancet Infect Dis. 2018 Dec;18(12):1350-1359. doi: 10.1016/S1473-3099(18)30496-1. Epub 2018 Oct 18. PMID 30342828
- [Background] Paris L, Magni R, Zaidi F, Araujo R, Saini N, Harpole M, Coronel J, Kirwan DE, Steinberg H, Gilman RH, Petricoin EF 3rd, Nisini R, Luchini A, Liotta L. Urine lipoarabinomannan glycan in HIV-negative patients with pulmonary tuberculosis correlates with disease severity. Sci Transl Med. 2017 Dec 13;9(420):eaal2807. doi: 10.1126/scitranslmed.aal2807. PMID 29237757
- [Background] Wood A, Barizuddin S, Darr CM, Mathai CJ, Ball A, Minch K, Somoskovi A, Hamasur B, Connelly JT, Weigl B, Andama A, Cattamanchi A, Gangopadhyay K, Bok S, Gangopadhyay S. Ultrasensitive detection of lipoarabinomannan with plasmonic grating biosensors in clinical samples of HIV negative patients with tuberculosis. PLoS One. 2019 Mar 26;14(3):e0214161. doi: 10.1371/journal.pone.0214161. eCollection 2019. PMID 30913250
- [Background] Nakhleh MK, Jeries R, Gharra A, Binder A, Broza YY, Pascoe M, Dheda K, Haick H. Detecting active pulmonary tuberculosis with a breath test using nanomaterial-based sensors. Eur Respir J. 2014 May;43(5):1522-5. doi: 10.1183/09031936.00019114. No abstract available. PMID 24789953
- [Background] Fernandez-Carballo BL, Broger T, Wyss R, Banaei N, Denkinger CM. Toward the Development of a Circulating Free DNA-Based In Vitro Diagnostic Test for Infectious Diseases: a Review of Evidence for Tuberculosis. J Clin Microbiol. 2019 Mar 28;57(4):e01234-18. doi: 10.1128/JCM.01234-18. Print 2019 Apr. PMID 30404942
- [Background] Ahmad Khan F, Pande T, Tessema B, Song R, Benedetti A, Pai M, Lonnroth K, Denkinger CM. Computer-aided reading of tuberculosis chest radiography: moving the research agenda forward to inform policy. Eur Respir J. 2017 Jul 13;50(1):1700953. doi: 10.1183/13993003.00953-2017. Print 2017 Jul. No abstract available. PMID 28705949
- [Background] Portevin D, Moukambi F, Clowes P, Bauer A, Chachage M, Ntinginya NE, Mfinanga E, Said K, Haraka F, Rachow A, Saathoff E, Mpina M, Jugheli L, Lwilla F, Marais BJ, Hoelscher M, Daubenberger C, Reither K, Geldmacher C. Assessment of the novel T-cell activation marker-tuberculosis assay for diagnosis of active tuberculosis in children: a prospective proof-of-concept study. Lancet Infect Dis. 2014 Oct;14(10):931-8. doi: 10.1016/S1473-3099(14)70884-9. Epub 2014 Aug 31. PMID 25185458
- [Background] Yoon C, Semitala FC, Atuhumuza E, Katende J, Mwebe S, Asege L, Armstrong DT, Andama AO, Dowdy DW, Davis JL, Huang L, Kamya M, Cattamanchi A. Point-of-care C-reactive protein-based tuberculosis screening for people living with HIV: a diagnostic accuracy study. Lancet Infect Dis. 2017 Dec;17(12):1285-1292. doi: 10.1016/S1473-3099(17)30488-7. Epub 2017 Aug 25. PMID 28847636
- [Background] Schmidt S. Bringing cheap and accurate tuberculosis tests to Africa. University of Wisconsin - News. 2018.
- [Background] Luabeya AK, Wood RC, Shenje J, Filander E, Ontong C, Mabwe S, Africa H, Nguyen FK, Olson A, Weigel KM, Jones-Engel L, Hatherill M, Cangelosi GA. Noninvasive Detection of Tuberculosis by Oral Swab Analysis. J Clin Microbiol. 2019 Feb 27;57(3):e01847-18. doi: 10.1128/JCM.01847-18. Print 2019 Mar. PMID 30541931
- [Background] Mesman AW, Calderon R, Soto M, Coit J, Aliaga J, Mendoza M, Franke MF. Mycobacterium tuberculosis detection from oral swabs with Xpert MTB/RIF ULTRA: a pilot study. BMC Res Notes. 2019 Jun 20;12(1):349. doi: 10.1186/s13104-019-4385-y. PMID 31221195
- [Background] Liu C, Lyon CJ, Bu Y, Deng Z, Walters E, Li Y, Zhang L, Hesseling AC, Graviss EA, Hu Y. Clinical Evaluation of a Blood Assay to Diagnose Paucibacillary Tuberculosis via Bacterial Antigens. Clin Chem. 2018 May;64(5):791-800. doi: 10.1373/clinchem.2017.273698. Epub 2018 Jan 18. PMID 29348166
- [Background] Walker TM, Kohl TA, Omar SV, Hedge J, Del Ojo Elias C, Bradley P, Iqbal Z, Feuerriegel S, Niehaus KE, Wilson DJ, Clifton DA, Kapatai G, Ip CLC, Bowden R, Drobniewski FA, Allix-Beguec C, Gaudin C, Parkhill J, Diel R, Supply P, Crook DW, Smith EG, Walker AS, Ismail N, Niemann S, Peto TEA; Modernizing Medical Microbiology (MMM) Informatics Group. Whole-genome sequencing for prediction of Mycobacterium tuberculosis drug susceptibility and resistance: a retrospective cohort study. Lancet Infect Dis. 2015 Oct;15(10):1193-1202. doi: 10.1016/S1473-3099(15)00062-6. Epub 2015 Jun 23. PMID 26116186
- [Background] Colman RE, Mace A, Seifert M, Hetzel J, Mshaiel H, Suresh A, Lemmer D, Engelthaler DM, Catanzaro DG, Young AG, Denkinger CM, Rodwell TC. Whole-genome and targeted sequencing of drug-resistant Mycobacterium tuberculosis on the iSeq100 and MiSeq: A performance, ease-of-use, and cost evaluation. PLoS Med. 2019 Apr 30;16(4):e1002794. doi: 10.1371/journal.pmed.1002794. eCollection 2019 Apr. PMID 31039166
- [Background] de Vos M, Ley SD, Wiggins KB, Derendinger B, Dippenaar A, Grobbelaar M, Reuter A, Dolby T, Burns S, Schito M, Engelthaler DM, Metcalfe J, Theron G, van Rie A, Posey J, Warren R, Cox H. Bedaquiline Microheteroresistance after Cessation of Tuberculosis Treatment. N Engl J Med. 2019 May 30;380(22):2178-2180. doi: 10.1056/NEJMc1815121. No abstract available. PMID 31141643
- [Background] Shin SS, Modongo C, Baik Y, Allender C, Lemmer D, Colman RE, Engelthaler DM, Warren RM, Zetola NM. Mixed Mycobacterium tuberculosis-Strain Infections Are Associated With Poor Treatment Outcomes Among Patients With Newly Diagnosed Tuberculosis, Independent of Pretreatment Heteroresistance. J Infect Dis. 2018 Nov 5;218(12):1974-1982. doi: 10.1093/infdis/jiy480. PMID 30085153
- [Background] Colman RE, Schupp JM, Hicks ND, Smith DE, Buchhagen JL, Valafar F, Crudu V, Romancenco E, Noroc E, Jackson L, Catanzaro DG, Rodwell TC, Catanzaro A, Keim P, Engelthaler DM. Detection of Low-Level Mixed-Population Drug Resistance in Mycobacterium tuberculosis Using High Fidelity Amplicon Sequencing. PLoS One. 2015 May 13;10(5):e0126626. doi: 10.1371/journal.pone.0126626. eCollection 2015. PMID 25970423
- [Background] Metcalfe JZ, Streicher E, Theron G, Colman RE, Penaloza R, Allender C, Lemmer D, Warren RM, Engelthaler DM. Mycobacterium tuberculosis Subculture Results in Loss of Potentially Clinically Relevant Heteroresistance. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e00888-17. doi: 10.1128/AAC.00888-17. Print 2017 Nov. PMID 28893776
- [Background] Lee JJ, Feng L. Randomized phase II designs in cancer clinical trials: current status and future directions. J Clin Oncol. 2005 Jul 1;23(19):4450-7. doi: 10.1200/JCO.2005.03.197. PMID 15994154
- [Background] Fleming TR. One-sample multiple testing procedure for phase II clinical trials. Biometrics. 1982 Mar;38(1):143-51. PMID 7082756
- [Derived] Crowder R, Thangakunam B, Andama A, Christopher DJ, Dalay V, Nwamba W, Kik SV, Van Nguyen D, Nhung NV, Phillips PPJ, Ruhwald M, Theron G, Worodria W, Yu C, Nahid P, Cattamanchi A, Gupta-Wright A, Denkinger CM. Diagnostic accuracy of TB screening tests in a prospective multinational cohort: Chest-X-ray with computer-aided detection, Xpert TB host response, and C-reactive protein. Clin Infect Dis. 2024 Nov 7:ciae549. doi: 10.1093/cid/ciae549. Online ahead of print. PMID 39509711
- [Derived] Crowder R, Thangakunam B, Andama A, Christopher DJ, Dalay V, Dube-Nwamba W, Kik SV, Nguyen DV, Nhung NV, Phillips PP, Ruhwald M, Theron G, Worodria W, Yu C, Nahid P, Cattamanchi A, Gupta-Wright A, Denkinger CM; R2D2 TB Network. Head-to-head comparison of diagnostic accuracy of TB screening tests: Chest-X-ray, Xpert TB host response, and C-reactive protein. medRxiv [Preprint]. 2024 Jun 21:2024.06.20.24308402. doi: 10.1101/2024.06.20.24308402. PMID 38947093
- [Derived] Gupta-Wright A, Ha H, Abdulgadar S, Crowder R, Emmanuel J, Mukwatamundu J, Marcelo D, Phillips PPJ, Christopher DJ, Nhung NV, Theron G, Yu C, Nahid P, Cattamanchi A, Worodria W, Denkinger CM; R2D2 TB Network. Evaluation of the Xpert MTB Host Response assay for the triage of patients with presumed pulmonary tuberculosis: a prospective diagnostic accuracy study in Viet Nam, India, the Philippines, Uganda, and South Africa. Lancet Glob Health. 2024 Feb;12(2):e226-e234. doi: 10.1016/S2214-109X(23)00541-7. PMID 38245113